CLINICAL TRIAL: NCT04995991
Title: Rhythmic Reading Training (RRT): Comparing the Rhythmic and Visual Contributions to Reading Improvement in Developmental Dyslexia
Brief Title: Rhythmic Reading Training: Comparing the Rhythmic and Visual Contributions to Reading Improvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); ASST Fatebenefratelli Sacco (Other); Associazione La Nostra Famiglia, Como, Italy (Unknown)
Responsible Party: Principal Investigator, Alice Cancer, Principal Investigator, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRT-VISUALCUE
Record Dates: First submitted 2021-07-16; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Developmental Dyslexia
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RRT rhythm only (Experimental): 10 RRT rhythm only sessions of 60 minutes, twice a week under the supervision of a trainer
  Interventions: Behavioral: RRT rhythm only
- RRT rhythm + visual cue (Experimental): 10 RRT rhythm + visual cue sessions of 60 minutes, twice a week under the supervision of a trainer
  Interventions: Behavioral: RRT rhythm + visual cue
- No intervention (No Intervention): 5 weeks no intervention period

INTERVENTIONS:
Behavioral: RRT rhythm only — RRT is a child-friendly computerized reading training program designed for Italian students with DD aged 8-14 yrs. The main feature of this intervention is the integration of a traditional remediation approach (sublexical treatment) with rhythm processing. Therefore, all reading exercises are characterized by a rhythmic accompaniment with gradually increasing speed. In this condition, the RRT activities comprise only a rhythm accompaniment and no visual cue.
  Arms: RRT rhythm only
Behavioral: RRT rhythm + visual cue — RRT is a child-friendly computerized reading training program designed for Italian students with DD aged 8-14 yrs. The main feature of this intervention is the integration of a traditional remediation approach (sublexical treatment) with rhythm processing. Therefore, all reading exercises are characterized by a rhythmic accompaniment with gradually increasing speed. In this condition, the rhythmic accompaniment is synchronize with a visual cue (the verbal stimuli are highlighted using a red font in synchrony with the rhythm).
  Arms: RRT rhythm + visual cue

SUMMARY:
The main objective of the study is to evaluate the specific effect of the sub-components of the reading training program Rhythmic Reading Training (RRT) on reading speed and accuracy in a sample of Italian students with developmental dyslexia (DD). More precisely, in order to better understand the neuropsychological mechanisms involved in reading improvements following RRT, the specific contribution of the visual component of the training (presence of a visual cue) will be investigated in a study with between-groups design.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with DD (ICD-10 code: F81.0) on the basis of standard inclusion and exclusion criteria (ICD-10: World Health Organization, 1992) and of the diagnosis procedure followed in the Italian practice

Exclusion Criteria:

* presence of comorbidity with other neuropsychiatric or psychopathological conditions
* having been involved in previous reading intervention programs in the previous 3 months

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Word reading speed - DDE-2 | 5 weeks
  Word reading speed in syllable / second
Word reading accuracy - DDE-2 | 5 weeks
  Word reading accuracy in n. of errors
Word reading speed - DDE-2 | 3 months
  Word reading speed in syllable / second
Word reading accuracy - DDE-2 | 3 months
  Word reading accuracy in n. of errors
Pseudo-word reading speed - DDE-2 | 5 weeks
  Pseudo-word reading speed in syllable / second
Pseudo-word reading accuracy - DDE-2 | 5 weeks
  Pseudo-word reading accuracy in n. of errors
Pseudo-word reading speed - DDE-2 | 3 months
  Pseudo-word reading speed in syllable / second
Pseudo-word reading accuracy - DDE-2 | 3 months
  Pseudo-word reading accuracy in n. of errors
Text reading speed - MT-3-Clinica Battery | 5 weeks
  Text reading speed in syllable / second
Text reading accuracy - MT-3-Clinica Battery | 5 weeks
  Text reading accuracy in n. of errors
Text reading speed - MT-3-Clinica Battery | 3 months
  Text reading speed in syllable / second
Text reading accuracy - MT-3-Clinica Battery | 3 months
  Text reading accuracy in n. of errors

SECONDARY OUTCOMES:
Phonemic awareness task (Judica et al., in press) | 5 weeks
  N. of errors in phonemic blending + n. of errors in phonemic elision
Phonemic awareness task (Judica et al., in press) | 3 months
  N. of errors in phonemic blending + n. of errors in phonemic elision
Digit span (Wechsler Intelligence Scale for Children-IV, WISC-IV) | 5 weeks
  Forward and backward digit span
Digit span (Wechsler Intelligence Scale for Children-IV, WISC-IV) | 3 months
  Forward and backward digit span
Rapid Automatized naming task - RAN (De Luca et al., 2005) | 5 weeks
  RAN speed in seconds
Rapid Automatized naming task - RAN (De Luca et al., 2005) | 3 months
  RAN speed in seconds
Selective Auditory attention task - NEPSY-II | 5 weeks
  N. of errors
Selective Auditory attention task - NEPSY-II | 3 months
  N. of errors
Rhythm reproduction task | 5 weeks
  n. of correctly reproduced rhythmic patterns
Rhythm reproduction task | 3 months
  n. of correctly reproduced rhythmic patterns

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided